CLINICAL TRIAL: NCT02567071
Title: Retablissement Du Microbiote Naturel Apres Naissance Par Cesarienne
Brief Title: Natural Microbiota Restoration After C-section Birth
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C14-70; 2015-A00586-43 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-09-15; First posted 2015-10-02 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Insufficient Intestinal Microbiota Diversity After C-section Birth
Keywords: C-section; Microbiota

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Experimental): 75 children born by planned C-section will be exposed to the perineal microbiota of their mothers through perineal impregnated swab.
  Interventions: Other: perineal impregnated swab
- Placebo Group (Placebo Comparator): 75 children born by planned C-section will be exposed to clean swab.
  Interventions: Other: clean swab
- Control Group (No Intervention): 75 children born vaginally.

INTERVENTIONS:
Other: perineal impregnated swab — After planned C-section birth, newborns will suck on previously impregnated swab by perineal and vaginal mother secretions.
  Arms: Intervention Group
Other: clean swab — After planned C-section birth, newborns will suck on clean swab.
  Arms: Placebo Group

SUMMARY:
The proportion of cesarean deliveries reached 30% of births in the US in 2008, while in the 1970s, it rarely reached 15%, as recommended by WHO. According to recent reports in some hospitals in China the use of cesarean section increased from 5% in the 1970s to over 60%. The use of C-section continues to grow in every countries of the world despite that current knowledge leads us to think that the vaginal birth, retained through millennia during mammalian evolution, guarantees the implementation of the best suited intestinal microbiota to build immunity and beneficial protective functions under the balanced mutual association between the host and its microbiota. Oral administration of a previously impregnated swab, by vaginal and maternal perineal secretions, following birth by planned C-section, would restore the normal development of the newborn intestinal microbiota mimicking exposure to these secretions during vaginal delivery.

The expected benefit is the establishment of a rich and diverse microbiota in individuals in the intervention group and by extension improving the overall health of these individuals.

ELIGIBILITY:
Inclusion Criteria:

* over the age of legal majority
* delivery by planned C-section at term or vaginal delivery at term
* registered at a social security service

Exclusion Criteria:

* HIV or other STD patients
* immunocompromised patients
* known streptococcus B carriers
* known vaginal or perineal herpes infections
* chronic disease patients (obesity, diabetes, IBD)
* IMC before pregnancy > 30 kg/m²
* antibiotic treatments one month before delivery
* emergency C-section
* Premature delivery (<37 amenorrhea weeks)
* hospitalized for more than one week before delivery
* known HVC infections
* for the newborns: every diagnosed anomaly
* patients who do not understand the research procedures or those that are institutionalized, or those unable to give informed consent
* patients deprived of ther liberty by legal or administrative decisions
* patients under an exclusion period from another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Diversity of the intestinal microbiota | 1 year
  Intestinal microbiota diversity will be evluated through metagenomics.

SECONDARY OUTCOMES:
Health status | 1 year
  Health status of the newborn will be evaluated through questionnaries.

CONTACTS AND LOCATIONS:
Overall Officials: Jacky Nizard, MD, PhD, Principal Investigator — APHP
Locations (1):
- Service de Gynécologie-Obstétrique, Groupe Hospitalier Pitié-Salpêtrière, Paris, France